CLINICAL TRIAL: NCT04878523
Title: Investigation of the Efficacies of Multi Berries Juice on Anti Oxidant Effect and Improvement of Skin Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 20-082-B
Record Dates: First submitted 2021-05-06; First posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Skin Condition; Anti Oxidative Stress
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo drink (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo drink
- multi berries juice (Experimental)
  Interventions: Dietary Supplement: multi berries juice

INTERVENTIONS:
Dietary Supplement: multi berries juice — Testing product
  Other Names: Sei Bella™ Pure Essence Whitening Multi-Berries Drink
  Arms: multi berries juice
Dietary Supplement: Placebo drink — Blank
  Arms: Placebo drink

SUMMARY:
To assess multi berries juice on anti-oxidant effect and skin condition improvement

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged above 20 years old

Exclusion Criteria:

* Subject who is not willing to participate in this study.
* Patients with diseases of the skin, liver, kidney.
* Subjects who have known cosmetic, drug or food allergies, difficulty in digestive tract absorption or disorder.
* Female who is pregnant or nursing or planning to become pregnant during the course of the study.
* Received facial laser therapy, chemical peeling or UV overexposure in the past 4 weeks.
* Constant drug use

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
The change of skin UV spots | Change from Baseline skin UV spots at 8 weeks
  VISIA Complexion Analysis System was utilized to measure skin UV spots. Units: arbitrary units
The change of skin melanin index | Change from Baseline skin melanin index at 8 weeks
  Soft Plus was utilized to measure skin melanin index. Units: arbitrary units
The change of blood SOD content | Change from Baseline SOD content at 8 weeks
  Venous blood was sampled to measure concentrations of SOD
The change of blood total antioxidant capacity (TAC) | Change from Baseline TAC at 8 weeks
  Venous blood was sampled to measure concentrations of TAC
The change of skin L* value | Change from Baseline L* value at 8 weeks
  Chroma Meter MM500 was utilized to measure skin L* value. Units: arbitrary units, 0-100
The change of skin spots | Change from Baseline skin spots at 8 weeks
  VISIA Complexion Analysis System was utilized to measure skin spots. Units: arbitrary units
The change of skin brown spots | Change from Baseline skin brown spots at 8 weeks
  VISIA Complexion Analysis System was utilized to measure skin brown spots. Units: arbitrary units

SECONDARY OUTCOMES:
The change of skin moisture | Change from Baseline skin moisture at 4 weeks
  Corneometer® CM825 was utilized to measure skin moisture. Units: arbitrary Corneometer® units 0-120
The change of skin a* value | Change from Baseline a* value at 8 weeks
  Chroma Meter MM500 was utilized to measure skin a* value. Units: arbitrary units
The change of skin elasticity | Change from Baseline skin elasticity at 8 weeks
  Soft Plus was utilized to measure skin elasticity. Units: arbitrary units
The change of skin wrinkles | Change from Baseline skin wrinkles at 8 weeks
  VISIA Complexion Analysis System was utilized to measure skin wrinkles. Units: arbitrary units
The change of skin texture | Change from Baseline skin texture at 8 weeks
  VISIA Complexion Analysis System was utilized to measure skin texture. Units: arbitrary units
The change of skin pores | Change from Baseline skin pores at 8 weeks
  VISIA Complexion Analysis System was utilized to measure skin pores. Units: arbitrary units
The change of skin collagen density | Change from Baseline skin collagen density at 8 weeks
  DermaLab® Series SkinLab Combo was utilized to measure skin collagen density. Units: arbitrary units

OTHER OUTCOMES:
The change of total cholesterol of blood | Change from Baseline total cholesterol at 8 weeks
  Venous blood was sampled to measure total cholesterol
The change of triglyceride of blood | Change from Baseline triglyceride at 8 weeks
  Venous blood was sampled to measure triglyceride
The change of SGOT of blood | Change from Baseline SGOT at 8 weeks
  Venous blood was sampled to measure SGOT
The change of SGPT of blood | Change from Baseline SGPT at 8 weeks
  Venous blood was sampled to measure SGPT
The change of BUN of blood | Change from Baseline BUN at 8 weeks
  Venous blood was sampled to measure BUN
The change of uric acid of blood | Change from Baseline uric acid at 8 weeks
  Venous blood was sampled to measure uric acid
The change of creatinine of blood | Change from Baseline creatinine at 8 weeks
  Venous blood was sampled to measure creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hua Liang, Principal Investigator — Chia Nan University of Pharmacy ＆ Science
Locations (1):
- Chia Nan University of Pharmacy & Science, Tainan, Taiwan